CLINICAL TRIAL: NCT02024243
Title: Tissue Oxygenation and miR-210 Role In Wound Healing
Brief Title: Role of Tissue Oxygenation and the miR-210 Gene In Wound Healing
Acronym: miR210
Status: Terminated | Type: Observational
Why Stopped: No funding available to continue
Sponsor: Chandan Sen (Other)
Responsible Party: Sponsor-Investigator, Chandan Sen, Professor, Indiana University
Organization: Indiana University (Other)
Other Study IDs: 1901906845
Record Dates: First submitted 2013-12-19; First posted 2013-12-31 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Non-Diabetic Patients; Wound Leg; Chronic Ulcer Leg/Foot
Keywords: Micro RNA; Wound; Chronic Venous Leg Ulcer; VLU; miR210; Indiana University Health Comprehensive Wound Center (CWC)
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — wound tissue biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Venous leg ulcers: Patients visiting the Indiana University Health Comprehensive Wound Center, with a chronic venous leg ulcer(s), who qualify based on the study inclusion and exclusion criteria, will be involved in a 14-week (98 days) longitudinal observational study. All subjects in this arm will have wound measurements, photographs for digital planimetry to measure wound area, and two 3 mm punch tissue biopsies of the same wound/ulcer (for OCT & infection) on days day 0, 14, and 28. Biopsies will not be taken if the wound has closed by day 14 or 28. Patient charts will be reviewed 98 days (14 weeks) after enrollment to determine the final status of the wound as healed or not-healed.

SUMMARY:
Hypothesis: Elevated miR210 in the epidermis (outer layer of skin) of ischemic human wound edge tissue (tissue that has a lack of blood flow to it) is associated with poor healing outcome in a setting of standard clinical care.

Aim of the study: To determine whether elevated miR-210 in the epidermis of ischemic human wound edge tissue is associated with poor healing outcome in a setting of standard clinical care.

This study will last 14 weeks. Adult patients, who are non-diabetic or tightly controlled diabetic, and, who have chronic venous leg ulcers that have been open/not healed for at least 12 weeks, will be enrolled in this study. Patients will be recruited from the Indiana University Health Comprehensive Wound Center (CWC). On days 0, 14 and 28, patients will have the following performed: measurements and photographs taken of their wound; TCOM (transcutaneous oxygen measurement) or ABI to measure the amount of oxygen in the wound tissue, if receiving a tissue biopsy; and two 3-mm punch biopsies from the same wound/ulcer. Biopsies will not be taken if the wound has closed by day 14 or day 28. Additionally, patients' medical records will be reviewed throughout the study for 98 days (14 weeks) after enrollment to determine the final status of the wound as healed or not-healed. ABI will be completed per study personnel at initial visit for all consented subjects to ensure subject eligibility (as listed TCOM<30 mmHg in exclusion criteria). If ABI's are unable to be obtained, TCOM will be performed.

There will be a total of 5 visits for this study (6 total visits for patients with open wounds on day 28 of the study). Visits will occur on days 0, 7, 14, 21,28.

DETAILED DESCRIPTION:
The study is designed as 28-day prospective longitudinal observational study including a 98 day (14 week) follow-up photography of the wound to test whether wounds open on day 28 have closed on week 14, or if they have remained chronically open.

On days 0, 14 and 28 after enrollment, wound images will be obtained. Wound photographs are a part of standard care when patients come to the Comprehensive Wound Center (CWC). Images do not include the part of body that could lead to identification of the participants. In addition, following standard of care, two biopsies will be taken - one biopsy will be used for laser capture microdissection (LCM) and immunohistochemistry studies, while the other will be used for determination of infection status using quantitative bacterial cultures and Scanning Electron Microscopy (SEM) imaging for biofilm phenotyping.

The following will be completed on days 0, 14 and 28:

1. Wound measurements - Photographs for digital planimetry to measure wound area.
2. Two Wound-edge biopsies (3mm) - following wound bed preparation with 1% lidocaine local anesthetic, as required, two punch biopsies (3 mm each) will be obtained from the wound-edge (the leading 3mm edge of the skin at the perimeter) of the same wound/ulcer.
3. Data Collection - the following information will be collected during the enrollment visit and updated at each visit (weekly - on days 0, 7, 14, 21, 28 and 98 (week 14) ), as necessary, and entered onto the data collection form: Age; Sex; Race/Ethnicity; Current medications; Transcutaneous oxygen measurement(TCOM) <30 mmHg or ABI < 0.8; Wound location & Etiology; Other associated illnesses; Wound care modality/treatment; and Nutritional status will be recorded as documented by albumin levels and chart records.

Healing outcome: Wound photography will be performed every 7 days (every week) as a part of the current standard of care. Based on wound measurements from days 0 and 28 , patients will be classified as either healing or non-healing, per criteria described in the study proposal/protocol.

There will be a total of 5 visits for this study (6 total visits for patients with open wounds on day 28 of the study). Visits will occur on days 0, 7, 14, 21 and 28.

ELIGIBILITY:
Inclusion Criteria:

* Ages 30 + years
* Presence of 1 or more non-neuropathic venous stasis leg ulcer(s) (VLU) confirmed by vascular duplex
* Chronic - Wound open >4 weeks

Exclusion Criteria:

* Individuals who are deemed unable to understand the procedures, risks, and benefits of the study (i.e., informed consent) will be excluded
* Pregnant women
* Diabetes with hemoglobin A1C > 9%
* Subjects with marked immunodeficiency (i.e., patients with HIV/AIDS, organ transplant, and/or cancer)
* Inadequate arterial supply, as evidenced by any of the following (for subjects receiving tissue biopsy with wounds below the knee):

  * TcOM < 30mmHg
  * ABI < 0.7 or >1.20
  * TBI < 0.6

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: non-diabetic or controlled diabetic, chronic (open >4 weeks) Venous leg ulcers
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Mean Change of miR210 Expression Across Healing Status (Healing vs. Non-Healing) | 28 Days
  The primary analysis will compare mean change cycle times (Delta Ct) of the baseline (d1) miR-210 expression across wound healing status (i.e., healing vs non-healing based on d28/d0 wound size (%) using either the two-sample t-test or the non-parametric Wilcoxon rank-sum test depending on the distribution of miR-210 and the homogeneity of the variance across groups.

CONTACTS AND LOCATIONS:
Overall Officials: Chandan K Sen, PhD, Principal Investigator — Indiana University Department of Surgery
Locations (3):
- United States (3):
  - Indiana University Health Comprehensive Wound Center, Indianapolis, Indiana
  - OSUWMC Comprehensive Wound Center (University Hospital East), Columbus, Ohio
  - OSUWMC Comprehensive Would Center (Martha Morehouse Medical Plaza), Columbus, Ohio

REFERENCES:
- See also: IU Department of Surgery — https://medicine.iu.edu/departments/surgery/
- See also: Indiana Center for Regenerative Medicine and Engineering — https://medicine.iu.edu/research/centers-institutes/regenerative-medicine-engineering/